CLINICAL TRIAL: NCT05965089
Title: A First-in-human, Randomised Double-blind, Placebo-controlled 2-part Study to Evaluate the Safety, Tolerability, Immunogenicity and Pharmacokinetics of Single Ascending Doses of AX-202 in Healthy Subjects and Multiple Ascending Doses of AX-202 in Patients With Mild to Moderate Chronic Plaque Psoriasis.
Brief Title: A First in Human Study of AX-202 in Healthy Subjects and Patients With Psoriasis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arxx Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AX-202-01
Record Dates: First submitted 2023-06-27; First posted 2023-07-28 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers; Mild to Moderate Psoriasis
Keywords: Single Ascending Doses; Multiple Ascending Doses; AX-202

STUDY DESIGN:
Intervention Model Description: Single-ascending doses in healthy subjects and multiple ascending doses in patients with mild to moderate chronic plaque psoriasis
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AX-202 (Experimental): Single and multiple ascending doses of AX-202
  Interventions: Biological: AX-202
- Placebo (Placebo Comparator): Single and multiple doses of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Placebo
  Arms: Placebo
Biological: AX-202 — Humanized monoclonal antibody
  Arms: AX-202

SUMMARY:
The first-in-human study will be performed in healthy volunteers and patients with a chronic inflammatory skin disease. The primary objective is to evaluate the safety, tolerability and pharmacokinetics of increasing doses of AX-202 infusion.

ELIGIBILITY:
Key Inclusion Criteria:

Part A / Single ascending doses:

* Male and female subjects must be between 18-55 years inclusive, at the time of informed consent.
* Subjects must have a Body Mass Index (BMI) ≥ 18 and ≤ 32 kg/m2 and weight of at least 45kg at screening.
* Subjects must be in good health as determined by medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory assessments at the time of screening, as judged by the Investigator.

Part B / Multiple ascending doses:

* Male and female patients must be between 18-65 years inclusive, at the time of informed consent.
* Patients must have a documented diagnosis of plaque psoriasis for ≥ 6 months prior to screening.
* Patients must have a Body Mass Index (BMI) ≥ 18 and ≤ 36 kg/m2 and weigh at least 45kg at screening.
* Patients must be in good health as determined by medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory assessments at the time of screening, as judged by the Investigator.

Key Exclusion Criteria:

Part A / Single ascending doses:

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the subject's safety during the clinical study or expose the subject to undue risk as judged by the Investigator.
* After a minimum of 10 minutes supine rest at the time of screening or on Day -1:

  * Systolic blood pressure <90 or >140 mmHg, or
  * Diastolic blood pressure <50 or >90 mmHg, or
  * Pulse <40 or >90 bpm
* Any clinically significant abnormalities in resting ECG at the time of screening or on Day -1 including prolonged QTcF (>450 ms for males; >470 ms for females using the mean of triplicate ECGs) and cardiac arrhythmias, as judged by the Investigator.
* Clinically significant abnormalities in renal function at screening.
* Clinically significant abnormalities in liver function at screening.
* Haemoglobin < 130 g/l for males or <120 g/l for females at screening.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP (Day 1).
* Malignancy within the past 5 years of screening with the exception of in situ removal of basal cell carcinoma or resected benign colonic polyps.
* Any planned major surgery within the duration of the study or in the 30 days following study completion.
* History of latent or active tuberculosis or a positive QuantiFERON® TB Gold test at screening.
* Females who are pregnant, breast feeding, lactating or plan to be pregnant during the study period or 120 days after.
* Female subjects with a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening or on Day -1.
* Positive serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV) 1 and/or 2 antibodies at screening.
* A Positive test for active COVID -19 prior to dosing on Day 1.
* History of any drug and/or alcohol abuse in the past 2 years prior to screening.
* Regular alcohol consumption of >14 units per week.
* Positive urine drugs of abuse test and/or alcohol breath test at screening or on admission to the unit on Day -1 that cannot be accounted for by concomitant medication in the opinion of the Investigator.
* Current or previous use of tobacco, nicotine products or e-cigarettes in the past 6 months.
* Smoking history of > 5 pack years.
* Positive urine cotinine test at screening or Day -1.
* Receiving any of the prohibited concomitant medications as specified in Section 5.5.3.1.
* Known history of intolerance or hypersensitivity to AX-202 or to any other component of the formulation.
* Known history of intolerance to placebo or excipients.
* Participation in another clinical study with an experimental drug within 3 months (non-biologic), 6 months (biologic) or 5 half-lives, whichever is longer, before the administration of IMP.

Part B / Multiple ascending doses:

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition other than psoriasis that could interfere with the patient's safety during the clinical study or expose the patient to undue risk as judged by the Investigator.
* A diagnosis of non-plaque psoriasis.
* Plaque psoriasis restricted to the scalp, palms, soles and face.
* Pustular, erythrodermic, inverse, and guttate psoriasis
* Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium)
* Diagnosis of psoriatic arthritis, uveitis, inflammatory bowel disease, or other immune-mediated conditions that are commonly associated with psoriasis for which a patient requires current systemic (oral, subcutaneous [SC], or IV) (including corticosteroids, immunosuppressants, biologics) immunosuppressant medical treatment.
* Presence of other skin conditions that could interfere with psoriasis evaluation or assessments as judged by the Investigator.
* After a minimum of 10 minutes supine rest at the time of screening or on Day -1:

  * Systolic blood pressure <90 or >140 mmHg, or
  * Diastolic blood pressure <50 or >90 mmHg, or
  * Pulse <40 or >90 bpm 9. Any clinically significant abnormalities in resting ECG at the time of screening or on Day -1 including prolonged QTcF (>450 ms for males; >470 ms for females using the mean of triplicate ECG's) and cardiac arrhythmias, as judged by the Investigator.
* Clinically significant abnormalities in renal function at screening.
* Clinically significant abnormalities in liver function at screening.
* Haemoglobin <130 g/l for males or <120 g/l for females at screening.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP (Day 1).
* Malignancy within the past 5 years of screening with the exception of in-situ removal of basal cell carcinoma or resected benign colonic polyps.
* Any planned major surgery within the duration of the study or in the 30 days following study completion.
* History of latent or active tuberculosis, or a positive QuantiFERON® TB Gold result at screening.
* Females who are pregnant, breast feeding, lactating or plan to be pregnant during the study period or 120 days after.
* Female patients with a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening or on Day -1.
* Positive serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV) 1 and/or 2 antibodies at screening.
* A Positive test for active COVID -19 prior to dosing on Day 1.
* History of any drug and/or alcohol abuse in the past 2 years prior to screening.
* Regular alcohol consumption of >14 units per week.
* Positive urine drugs of abuse test and/or alcohol breath test at screening or on admission to the unit on Day -1 that cannot be accounted for by concomitant medication in the opinion of the Investigator.
* Receiving any of the prohibited concomitant medications as specified in Section 5.5.3.2.
* Any clinically significant infection requiring antimicrobial treatment in the 2 weeks prior to Day 1.
* Known history of intolerance or hypersensitivity to AX-202 or to any other component of the formulation.
* Known history of intolerance to placebo or excipients.
* Participation in another clinical study with an experimental drug within 3 months (non-biologic), 6 months (biologic) or 5 half-lives, whichever is longer, before the administration of IMP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of a single ascending IV dose of AX-202 in healthy subjects and multiple ascending IV doses of AX-202 in patients with mild to moderate chronic plaque psoriasis by monitoring of adverse events. | Until 100 days after last dose
  Number of patients with AE's
To assess the safety and tolerability of a single ascending IV dose of AX-202 in healthy subjects and multiple ascending IV doses of AX-202 in patients with mild to moderate chronic plaque psoriasis by physical examinations. | Until 100 days after last dose
  Number of patients with clinically significant findings on physical examinations
To assess the safety and tolerability of a single ascending IV dose of AX-202 in healthy subjects and multiple ascending IV doses of AX-202 in patients with mild to moderate chronic plaque psoriasis by assessment of infusion related reactions | Until 100 days after last dose
  Number of patients with infusion related reactions
To assess the safety and tolerability of a single ascending IV dose of AX-202 in healthy subjects and multiple ascending IV doses of AX-202 in patients with mild to moderate chronic plaque psoriasis by monitoring of vital signs | Until 100 days after last dose
  Number of patients with clinically significant changes from baseline in vital signs
To assess the safety and tolerability of a single ascending IV dose of AX-202 in healthy subjects and multiple ascending IV doses of AX-202 in patients with mild to moderate chronic plaque psoriasis by monitoring of clinical laboratory parameters | Until 100 days after last dose
  Number of patients with clinically significant change from baseline in clinical laboratory test results.
To assess the safety and tolerability of a single ascending IV dose of AX-202 in healthy subjects and multiple ascending IV doses of AX-202 in patients with mild to moderate chronic plaque psoriasis by ECG monitoring | Until 100 days after last dose
  Number of patients with clinically significant change from baseline in ECG parameters

SECONDARY OUTCOMES:
To characterise systemic PK of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Calculation of maximum serum concentration (Cmax) of AX-202
To characterise systemic PK of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Calculation of time to maximum concentration (tmax) of AX-202
To characterise systemic PK of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Calculation of the area under the plasma concentration-time curve (AUC)
To characterise systemic PK of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Calculation of the half-life of AX-202
To characterise systemic PK of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Calculation of the clearance (CL) of AX-202
To characterise systemic PK of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Calculation of volume of distribution at steady state (Vss)
To evaluate immunogenicity of AX-202 after a single ascending IV dose in healthy subjects and after multiple ascending IV doses in patients with mild to moderate chronic plaque psoriasis. | Until 100 days after last dose
  Number of participants with anti-drug antibodies against AX-202

CONTACTS AND LOCATIONS:
Locations (1):
- Medicines Evaluation Unit, Manchester, Wythenshawe, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analysed during the current study will be available upon request from Arxx Therapeutics, contact details can be found at the following website: https://arxxtx.com/.
  Deidentified individual participant data will be available after the study has been reported, approximately 12 months after the study's concluded. These data will be available for 36 months. These data will be shared with Investigators whose proposed use of the data has been approved by Arxx Therapeutics. Proposals may be submitted up to 36 months following reporting of the study.
Time Frame: Deidentified data will be available approximately 12 months after the study's concluded. These data will be available for 36 months. Proposals for use of data may be submitted up to 36 months following reporting of the study.
Access Criteria: Data will be shared with Investigators whose proposed use of the data has been approved by Arxx Therapeutics.

REFERENCES:
- [Derived] Borchert SV, Hallen J, Hussain RI, Holyer I, Troelsen JT, Klingelhofer J. Development of CAL101-a humanized monoclonal antibody targeting S100A4 to inhibit proinflammatory and profibrotic signaling. J Pharmacol Exp Ther. 2025 Nov;392(11):103722. doi: 10.1016/j.jpet.2025.103722. Epub 2025 Sep 24. PMID 41124966